CLINICAL TRIAL: NCT01197092
Title: A Study Evaluating the Effects of a Regenerative Mitochondrial Medication on Physiological Parameters in Case of Diabetes Mellitus Type II
Brief Title: The Effects of a Regenerative Mitochondrial Medication on Physiological Parameters in Case of Diabetes Mellitus Type II
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Center for Integrative Medicine, Germany (Other)
Responsible Party: Rainer Mutschler, Center for Integrative Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CS-101-01
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-09

CONDITIONS: Diabetes Mellitus, Type II
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Home Infusion Therapy; Nutrition Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Verum (Active Comparator)
  Interventions: Dietary Supplement: Mitochondrial preparations; Dietary Supplement: Infusion therapy; Device: Webermedical device; Behavioral: Nutritional therapy
- Control (Experimental)
  Interventions: Behavioral: Nutritional therapy

INTERVENTIONS:
Dietary Supplement: Mitochondrial preparations — Oral therapy with mitochondrial preparations based on recipes of Dr Kremer and the Tisso company:
  ProEMSan (large intestinal symbionts with 31 strains of bacteria) Pro Basan (small intestinal symbionts) ProSirtusan (Polyphenol-mix and vitamins) ProVita D3 (Vitamin D3 supplement) ProOmega (Omega 3-fatty acid preparation) ProCarnitin (Carnitine-preparation) ProSango Vital (trace element preparation)
  Arms: Verum
Dietary Supplement: Infusion therapy — Infusion therapy in the form of a complex mix: 500ml-solution with trace elements, amino acids and antioxidants.
  Arms: Verum
Device: Webermedical device — Intravenous-Blood-Laser-Therapy: the Webermedical device will be used
  Arms: Verum
Behavioral: Nutritional therapy — Nutritional therapy based on IgG-blood results. Significant antibody-formation against foodstuffs will be ascertained (in foodstuffs evaluated through the BioMedicalScreen), will be taken out of the diet - the background being the additional lowering of risk potential of those antibodies causing the so called "silent inflammation" (sub-clinical inflammation) -ultimately an anti-inflammatory diet will be given in the protocol. The following have special focus: gluten, cow's milk, fish, meat, nuts.

SUMMARY:
A treatment with the concept of mitochondrial medication developed by Dr Heinrich Kremer can demonstrably improve and successfully treat actual parameters of Diabetes Mellitus II as well as its risk factors.

ELIGIBILITY:
Inclusion Criteria:

* men and women between the ages of 18 and 60
* recently diagnosed Diabetes Type II (within the last 12 months)

Exclusion Criteria:

* no orally-taken medication up to present
* no insulin therapy
* no diseases resulting from diabetes like Nephropathy, Neuropathy, Angiopathy or Retinopathy
* fasting blood sugar values in the morning under 200mmol
* sufficient production of insulin

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
HbA1c Test (Glycated hemoglobin) | 4 month average
  Laboratory test

SECONDARY OUTCOMES:
Blood count | 4 month average
  Laboratory test
Electrolytes | 4 month average
  Laboratory test
Liver, pancreatic and kidney retention values | 4 month average
  Laboratory test
Lipids: Cholesterol,Triglycerides | 4 month average
  Laboratory test
Oxyd LDL (low-density lipoprotein cholesterol) | 4 month average
  Laboratory test
Free lipids fasting | 4 month average
  Laboratory test
Lipoprotein A | 4 month average
  Laboratory test
Fibrinogen | 4 month average
  Laboratory test
CRP (C Reactive protein) | 4 month average
  Laboratory test
LDH-Isoenzymes (Lactate dehydrogenase) | 4 month average
  Laboratory test
Homocysteins | 4 month average
  Laboratory test
Nutrient IgGs Panels (BiomedicalScreen) | 4 month average
  Laboratory test
Insulin, Adiponectin, Leptin | 4 month average
  Laboratory test
Potassium, selene, magnesium, zinc in whole blood | 4 month average
  Laboratory test
SHbG, full-testosterone (Androgen-Index) | 4 month average
  Laboratory test
PlasminInhibitor I | 4 month average
  Laboratory test
Vitamins B1,B2,B6,B 12, Vitamin D | 4 month average
  Laboratory test

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Mutschler, MD, Principal Investigator
Locations (1):
- CFI Centrum für Integrative Medizin, Speyer, Germany